CLINICAL TRIAL: NCT01757301
Title: Comprehensive vs. Assisted Management of Mood and Pain Symptoms (CAMMPS) Trial
Brief Title: Comprehensive vs. Assisted Management of Mood and Pain Symptoms
Acronym: CAMMPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIR 12-095
Record Dates: First submitted 2012-12-20; First posted 2012-12-28 (Estimated); Results first posted 2019-03-13 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Pain; Depression; Anxiety; Musculoskeletal; Fibromyalgia
Keywords: Pain; Depression; Anxiety; Musculoskeletal; Fibromyalgia
MeSH Terms: conditions — Pain; Depression; Anxiety Disorders; Fibromyalgia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Assisted Symptom Management (ASM) (Active Comparator): There will be 2 principal components to assisted symptom management (ASM): automated symptom monitoring, along with pain and mood self-management modules.
  Interventions: Other: Assisted Symptom Management (ASM)
- Comprehensive Symptom Management (CSM) (Experimental): This arm couples ASM with care management by a nurse-physician team, thus testing "combined" therapy vs. "monotherapy" (ASM only).
  Interventions: Other: Comprehensive Symptom Management (CSM)

INTERVENTIONS:
Other: Assisted Symptom Management (ASM) — There will be 2 principal components to assisted symptom management (ASM): automated symptom monitoring, along with pain and mood self-management modules.
  Arms: Assisted Symptom Management (ASM)
Other: Comprehensive Symptom Management (CSM) — This arm couples ASM with care management by a nurse-physician team, thus testing "combined" therapy vs. "monotherapy" (ASM only).
  Arms: Comprehensive Symptom Management (CSM)

SUMMARY:
Pain is the most common presenting symptom in medical outpatients, and depression and anxiety are the two most common mental disorders. All three conditions are often inadequately treated and result in substantial disability, reduced health-related quality of life, and increased health care costs and utilization. Additionally, pain, anxiety, and depression (PAD) are frequently comorbid with one another and have reciprocal negative effects on treatment response and additive effects on adverse health outcomes. The PAD triad is especially burdensome in Veterans, with their high prevalence of chronic pain, depression, PTSD, and other anxiety disorders. The Comprehensive vs. Assisted Management of Mood and Physical Symptoms (CAMMPS) study is a randomized comparative effectiveness trial designed to test the relative effectiveness of a lower-resource vs. a higher-resource enhancement of usual primary care in the management of Veterans suffering from with pain plus comorbid anxiety and/or depression.

DETAILED DESCRIPTION:
The Comprehensive vs. Assisted Management of Mood and Physical Symptoms (CAMMPS) study is a randomized comparative effectiveness trial designed to test the relative effectiveness of a lower-resource vs. a higher-resource enhancement of usual primary care in the management of Veterans suffering from with pain plus comorbid anxiety and/or depression.

This is a single-site study enrolling Veterans. Patients followed in primary care clinics at the Roudebush VAMC will be eligible if they have clinically significant levels of pain plus comorbid anxiety and/or depression. A total of 300 eligible patients who provide informed consent will be randomized to one of two treatment arms. One group (n=150) will receive assisted symptom management (ASM) consisting of automated symptom monitoring by interactive voice recording or Internet and prompted pain self-management guided by symptom levels. The second group (n=150) will receive comprehensive symptom management (CSM) which combines ASM with optimized medication management delivered by a nurse-physician specialist team and facilitated mental health care. This team will partner with both VA primary care physicians and psychologists embedded in primary care to monitor and adjust treatments using evidence-based analgesic and antidepressant algorithms, reinforced self-management, and care coordination. The investigators postulate that although both interventions are likely to be beneficial, CSM will be superior to ASM.

In short, this trial compares: 1) usual care plus assisted symptom management (ASM) vs. 2) usual care plus ASM plus optimized medication and care management and facilitated mental health care (CSM). Outcomes will be assessed at baseline, 1, 3, 6, and 12 months. The primary outcome is a composite pain-anxiety-depression severity score. Secondary outcomes include individual pain, anxiety, and depression scores; functional status and health-related quality of life; treatment satisfaction; and perceived barriers and facilitators of the CSM and ASM interventions. The rationale for ASM is preliminary evidence of its effectiveness and its lower use of resources. The rationale for CSM is that the addition of optimized medication management, facilitated mental health care, and coordination with both primary care physicians/Patient Aligned Care Teams (PACTs) and psychologists for the PAD symptoms should substantially enhance the benefits of ASM.

ELIGIBILITY:
Inclusion Criteria:

Individuals must be patients of the Richard L. Roudebush VAMC in Indianapolis, Indiana Individuals will be eligible if they have pain plus comorbid anxiety and/or depression.

* Pain must:

  * be musculoskeletal, either localized (in the arms, legs, back, or neck) or widespread (fibromyalgia)
  * have persisted 3 months or longer despite a trial of at least one analgesic medication
  * at least moderate in severity, defined as a Brief Pain Inventory average severity score of 5 or greater
* Depression must be of at least moderate severity, defined as a PHQ-8 score of 10 or greater with either depressed mood and/or anhedonia being endorsed, OR
* Anxiety must be of at least moderate severity, defined as a GAD-7 score of 10 or greater, OR
* A composite mood score (anxiety and depression) of sufficient severity, defined as a GAD-7 + PHQ-8 score of 12 or greater.

Exclusion Criteria:

Individuals will be excluded if they:

* do not speak English
* have moderately severe cognitive impairment as defined by a validated 6-item cognitive screener
* have schizophrenia, bipolar disorder or other psychosis
* have other severe mental illness and/or high risk of suicide
* are pregnant
* have an anticipated life expectancy of less than 12 months. Patients who are on antidepressants but still meet the PHQ-9 and/or GAD-7 entry criterion for clinical depression and/or anxiety may still be eligible if they have been on an adequate dose of the antidepressant for an adequate duration of time (i.e., 12 weeks).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 296 (Actual)
Dates: Start 2014-01-02 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kurt Kroenke, MD, Principal Investigator — Richard L. Roudebush VA Medical Center, Indianapolis, IN
Locations (1):
- Richard L. Roudebush VA Medical Center, Indianapolis, IN, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Toussaint A, Kroenke K, Baye F, Lourens S. Comparing the Patient Health Questionnaire - 15 and the Somatic Symptom Scale - 8 as measures of somatic symptom burden. J Psychosom Res. 2017 Oct;101:44-50. doi: 10.1016/j.jpsychores.2017.08.002. Epub 2017 Aug 2. PMID 28867423
- [Background] Kroenke K, Evans E, Weitlauf S, McCalley S, Porter B, Williams T, Baye F, Lourens SG, Matthias MS, Bair MJ. Comprehensive vs. Assisted Management of Mood and Pain Symptoms (CAMMPS) trial: Study design and sample characteristics. Contemp Clin Trials. 2018 Jan;64:179-187. doi: 10.1016/j.cct.2017.10.006. Epub 2017 Oct 12. PMID 29031492

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two participants were excluded from the study after enrollment. Both participants failed screening and were considered ineligible.
Period: Overall Study
Arm/Group | Assisted Symptom Management (ASM) | Comprehensive Symptom Management (CSM)
Started | 147 | 147
Completed | 134 | 133
Not Completed | 13 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Assisted Symptom Management (ASM) | Comprehensive Symptom Management (CSM) | Total
Number analyzed (Participants) | 147 | 147 | 294
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.9 (11.7) | 56.9 (12.5) | 57.4 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 23 | 37
  Male | 133 | 124 | 257
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 24 | 21 | 45
  White | 117 | 116 | 233
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 7 | 13
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 147 | 147 | 294

OUTCOME MEASURES:

1. Primary Outcome: Composite Z-score of Pain-anxiety-depression Severity
Description: The primary outcome measure is the composite z-score of the main pain, anxiety, and depression measures in this trial: the BPI, GAD-7, PHQ-9, respectively. A standard z-score is calculated for each scale as follows: subject's scale score minus the sample mean divided by the sample standard deviation. A composite pain-anxiety-depression score is the average of the standard z-scores for the 3 scales. This is a scale of effect size where 0 represents no change from baseline, and a negative number means improvement and a positive number means worsening. Each unit means one standard deviation change from the group at baseline. Practical minimum value= -2.0, maximum value= +2.0. Positive number indicates greater symptoms severity/worse outcomes.
Time Frame: 12 months
Population: Seven participants in the CSM group and seven participants in the ASM group had no follow-up assessments after baseline and were therefore not included in the primary MMRM analysis since at least one follow-up data point is required for MMRM.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Assisted Symptom Management (ASM): There will be 2 principal components to assisted symptom management (ASM): automated symptom monitoring, along with pain and mood self-management modules. Assisted Symptom Management (ASM): There will be 2 principal components to assisted symptom management (ASM): automated symptom monitoring, along with pain and mood self-management modules.
- Comprehensive Symptom Management (CSM): This arm couples ASM with care management by a nurse physician team, thus testing "combined" therapy vs.
  "monotherapy" (ASM only). Comprehensive Symptom Management (CSM): This arm couples ASM with care management by a nurse physician team, thus testing "combined" therapy vs. "monotherapy" (ASM only).
Arm/Group | Assisted Symptom Management (ASM) | Comprehensive Symptom Management (CSM)
Number analyzed (Participants) | 140 | 140
units on a scale | -0.52 (1.05) | -0.65 (0.94)

2. Secondary Outcome: Pain Average/Enjoyment of Life/General Activities Pain Scale (PEG)
Description: The PEG is a 3-item validated version of the Brief Pain Inventory. Minimum value = 0; maximum value = 10. Higher scores indicate greater symptom severity/worse outcomes.
Time Frame: 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Assisted Symptom Management (ASM) | Comprehensive Symptom Management (CSM)
Number analyzed (Participants) | 140 | 140
units on a scale | 6.0 (1.9) | 6.1 (2.0)

3. Secondary Outcome: Patient Health Questionnaire 9-item Depression Scale (PHQ-9)
Description: The PHQ-9 has been used in hundreds of research studies as a depression severity and outcome measure and, now translated into more than 80 languages, is among the most widely used depression measures in clinical practice. Minimum value = 0; maximum value = 27. Higher scores indicate greater symptom severity/worse outcomes.
Time Frame: 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Assisted Symptom Management (ASM) | Comprehensive Symptom Management (CSM)
Number analyzed (Participants) | 140 | 140
units on a scale | 11.4 (5.9) | 10.3 (5.3)

4. Secondary Outcome: Generalized Anxiety Disorder 7-Item Anxiety Scale (GAD-7)
Description: The GAD-7 is an anxiety severity measure, validated in several thousand primary care patients and increasingly used in clinical research and practice. It is also a good first-line measure for estimating the probability of 4 common anxiety disorders in primary care - generalized anxiety disorder, panic disorder, post-traumatic stress disorder, and social anxiety disorder. Minimum value = 0; maximum value = 21. Higher scores indicate greater symptom severity/worse outcomes.
Time Frame: 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Assisted Symptom Management (ASM) | Comprehensive Symptom Management (CSM)
Number analyzed (Participants) | 140 | 140
units on a scale | 8.4 (6.2) | 7.5 (5.4)

5. Secondary Outcome: Brief Pain Inventory (BPI)
Description: The BPI rates the intensity of pain on 4 items (current, worst, least, and average pain in past week), and the interference in 7 areas (mood, physical activity, work, social activity, relations with others, sleep, enjoyment of life). Minimum value = 0; maximum value = 10. Higher scores indicate greater symptom severity/worse outcomes.
Time Frame: 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Assisted Symptom Management (ASM) | Comprehensive Symptom Management (CSM)
Number analyzed (Participants) | 140 | 140
units on a scale | 5.0 (2.3) | 5.0 (2.2)

ADVERSE EVENTS:
Time Frame: SAEs and AEs were assessed for each participant from baseline date through the date the 12 month interview was completed or through the date the participant withdrew participation (if applicable). The average timeframe among all participants was 365 days.
Description: SAEs were solicited and documented from all participants during 6 and 12 month outcome interviews and if spontaneously reported by participants. SAE/AEs were additionally solicited and documented from CSM participants during automated symptom monitoring, multiple nurse care manager phone calls and were documented when the nurse found evidence of an SAE/AE in a CSM participant's medical record. This method led to a much greater identification rate of AEs in CSM than in ASM participants.
Arm/Group | Assisted Symptom Management (ASM) | Comprehensive Symptom Management (CSM)
All-Cause Mortality (participants affected / at risk) | 1/147 | 2/147
Serious Adverse Events (participants affected / at risk) | 18/147 | 30/147
Other Adverse Events (participants affected / at risk) | 13/147 | 72/147
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Assisted Symptom Management (ASM) (N=147) | Comprehensive Symptom Management (CSM) (N=147)
Endorsed Suicidal Thoughts (Psychiatric disorders) | 1 (1) | 0 (0)
Hospitalization for Suicidal Behavior (Psychiatric disorders) | 0 (0) | 4 (4)
Hospitalization for pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Hospitalization for Influenza (General disorders) | 1 (1) | 0 (0)
Hospitalization for kidney stone (Renal and urinary disorders) | 1 (1) | 0 (0)
Broken kneecap (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Kneecap broken after falling on ice. Received urgent treatment at local hospital and scheduled surgery to repair.
Hospitalization for TIA (Nervous system disorders) | 1 (1) | 1 (1)
Hospitalization for wound (Infections and infestations) | 1 (1) | 3 (4)
Hospitalization for planned knee replacement (Surgical and medical procedures) | 1 (1) | 0 (0)
Hospitalization for planned angioplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Hospitalization for heart catheterization (Cardiac disorders) | 2 (2) | 0 (0)
Hospitalization for thyroidectomy (Endocrine disorders) | 1 (1) | 0 (0)
Hospitalization for planned hip surgery (Surgical and medical procedures) | 1 (1) | 1 (1)
Hospitalization for planned hernia repair (Surgical and medical procedures) | 2 (2) | 1 (1)
Hospitalization following emergency appendectomy (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hospitalization for diverticulitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Hospitalization for gastroparesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hospitalization for planned autologous fascial sling surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Diagnosis of Hodgkins Lymphoma (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Diagnosis made by GI following biopsy of lymph node during endoscopic ultrasound procedure.
Hospitalization following fall from ladder (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Hospitalized for pain control following fall from 10 foot ladder. Suffered several broken ribs.
ER visit for atypical chest pain (Cardiac disorders) | 0 (0) | 2 (2) — Presented to ER with atypical chest pain. Normal evaluation and work up. Released in stable condition.
Hospitalization for planned septoplasty (Surgical and medical procedures) | 0 (0) | 2 (2)
Hospitalization for substance abuse (General disorders) | 0 (0) | 3 (3)
Hospitalization following renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Diagnosis of deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
ER visit for fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Yearly surveillance for known prostate cancer (Renal and urinary disorders) | 0 (0) | 1 (1)
ER visit for trouble breathing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Surgery following dog attack injuries (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hospitalization for heart stent placement (Cardiac disorders) | 0 (0) | 1 (1)
Hospitalization following elective laminectomy/fusion (Surgical and medical procedures) | 0 (0) | 1 (1)
Hospitalization for polycythemia likely secondary to renal mass (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hospitalization for pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hospitalization for infection (Blood and lymphatic system disorders) | 1 (2) | 1 (1)
Hospitalized following stem cell transplant (Surgical and medical procedures) | 0 (0) | 1 (1)
Hospitalization for COPD (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Hospitalization for bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hospitalization for pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hospitalization for atypical chest pain (General disorders) | 0 (0) | 1 (1)
Hospitalization for collapsed lung (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hospitalization following amputation of left leg (Infections and infestations) | 1 (1) | 0 (0) — Participant had calcaneus removed which resulted in a bone infection. Left leg amputated as a result.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Assisted Symptom Management (ASM) (N=147) | Comprehensive Symptom Management (CSM) (N=147)
Triggered Suicidal Ideation Screener (Psychiatric disorders) | 13 (17) | 16 (23) — Responses were recorded as Adverse Events when participants responded Somewhat/Very Likely, or refused to answer how likely they were to act on their self-harm thoughts and/or if they reported nothing/no one to prevent them from self-harm.
Known medication side effects (General disorders) | 0 (0) | 61 (92)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-11-30): https://cdn.clinicaltrials.gov/large-docs/01/NCT01757301/Prot_SAP_000.pdf